CLINICAL TRIAL: NCT06183788
Title: Antibody-mediated NMDA Receptor Encephalitis: Symptoms, Biomarkers, and Mechanisms of the Prolonged Recovery Stage
Acronym: AMENDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Collaborators: Hospital Sant Joan de Deu (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HR22-00221
Record Dates: First submitted 2023-05-19; First posted 2023-12-28 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Anti-NMDA Receptor Encephalitis
Keywords: Cognitive Impairment; Encephalitis; Autoimmune; Cognitive rehabilitation
MeSH Terms: conditions — Anti-N-Methyl-D-Aspartate Receptor Encephalitis; Cognitive Dysfunction; Encephalitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-NMDARe patients with remote cognitive rehabilitation (Experimental): Participants of a prospective cohort in post-acute phase of the Antibody-mediated NMDA Receptor Encephalitis that will received a behavioral treatment.
  Interventions: Behavioral: Remote cognitive rehabilitation program

INTERVENTIONS:
Behavioral: Remote cognitive rehabilitation program — Remote cognitive rehabilitation program will be performed through an online validated platform (Guttmann NeuroPersonalTrainer: https://gnpt.es/) run by the psychologists team. This is a Sanitary Product with CE certification (Sanitary Product RPS/430/2014; International Patent [PCT/ES2008/00677]) and here will be used within its approved indications. The rehabilitation program will increase in difficulty and decrease in frequency during the first year of follow-up (V1-V3).

SUMMARY:
The encephalitis mediated by antibodies against the NMDA receptor (NMDARe) predominantly affects young adults and children resulting in severe neurologic and psychiatric deficits. After overcoming the acute stage, patients are left with long-lasting behavioral, cognitive, and psychiatric alterations with important socio-family-economical implications. Here investigators postulate that a better knowledge of this stage will improve treatment decisions and outcome.

In Aim 1, the post-acute stage will be clinically characterized, tools to remotely follow cognitive, behavioral and psychiatric deficits will be provided, and the impact of cognitive rehabilitation will be assessed.

In Aim 2, biomarkers (autoimmune, inflammatory, neuronal injury) will be identified as signatures of the acute and post-acute stages.

In Aim 3, a mouse model of NMDARe will be used to determine the underlying mechanisms and treatment of the postacute stage.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥12 years old with NMDARe in the post-acute stage of the disease;
* ≤6 months from hospital discharge (acute phase)

Exclusion Criteria (one of the following):

* Inability to obtain informed consent;
* inability to travel to the center.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Age | 18 months
  Age measured in years
Gender | 18 months
  Male or female
Vision condition | 18 months
  Studied by optometer
Handedness | 18 months
  Right- or Left-handed
General medical history | 18 months
  Description of the most important issues compiled in the general medical history of the participant
Allergies | 18 months
  List of allergies of each participant
Symptoms related to NMDARe | 18 months
  Detailed description of symptoms experienced before, during and after the post-acute phase of NMDARe.
Treatments | 18 months
  All treatments in which the participant is being involved.
Functional status | 18 months
  Functional status according to Modified Rankin Scale (mRS)
  Modified Rankin Scale:
  - Range: from 0 points (no symptoms) to 6 points (dead).
Intelligence Quotient | 18 months
  Estimated through General Ability Index (GAI; from Weschler Adult Intelligence Scale - IV (WAIS-IV).
  This index is obtained through Verbal Comprehension Index (VCI) and Perceptual Reasoning Index (PRI).
  * Range of GAI: from 40 to 160. Higher is better.
  * Range of VCI: from 50 to 150. Higher is better.
  * Range of PRI: from 50 to 150. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Verbal working memory | 18 months
  Verbal Working Memory: Working Memory Index (WMI) from WAIS-IV.
  - Range of WMI: from 50 to 150. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Phonological loop | 18 months
  Assessed by Forward order span of Digit span subtest from WAIS-IV.
  - Range: from 0 to 9
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Visual working memory | 18 months
  Visual Working Memory: Spatial location subtest from Weschler Memory Scale - IV (WMS-IV).
  - Range of Spatial Location subtest: from 0 to 32. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Verbal learning | 18 months
  Assessed by:
  Adults: España - Complutense Auditory-Verbal Learning Test (Test de Aprendizaje Verbal España - Complutense; TAVEC); or Infants: España - Complutense Auditory-Verbal Learning Test for Children (Test de Aprendizaje Verbal España - Complutense Infantil; TAVECI)
  - Total learning: range: from 0 to 80. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Proactive interference verbal memory | 18 months
  Assessed by:
  Adults: España - Complutense Auditory-Verbal Learning Test (Test de Aprendizaje Verbal España - Complutense; TAVEC); or Infants: España - Complutense Auditory-Verbal Learning Test for Children (Test de Aprendizaje Verbal España - Complutense Infantil; TAVECI)
  - Interference list: range: 0 to 15. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Short-term verbal memory | 18 months
  Assessed by:
  Adults: España - Complutense Auditory-Verbal Learning Test (Test de Aprendizaje Verbal España - Complutense; TAVEC); or Infants: España - Complutense Auditory-Verbal Learning Test for Children (Test de Aprendizaje Verbal España - Complutense Infantil; TAVECI)
  - Short-term memory free recall: range: 0 to 15. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Long-term verbal memory | 18 months
  Assessed by:
  Adults: España - Complutense Auditory-Verbal Learning Test (Test de Aprendizaje Verbal España - Complutense; TAVEC); or Infants: España - Complutense Auditory-Verbal Learning Test for Children (Test de Aprendizaje Verbal España - Complutense Infantil; TAVECI)
  - Long-term memory free recall: range: 0 to 15. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Verbal recognition memory | 18 months
  Assessed by:
  Adults: España - Complutense Auditory-Verbal Learning Test (Test de Aprendizaje Verbal España - Complutense; TAVEC); or Infants: España - Complutense Auditory-Verbal Learning Test for Children (Test de Aprendizaje Verbal España - Complutense Infantil; TAVECI)
  - Word-list Recognition: range: 0 to 15. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Verbal discrimination memory | 18 months
  Assessed by:
  Adults: España - Complutense Auditory-Verbal Learning Test (Test de Aprendizaje Verbal España - Complutense; TAVEC); or Infants: España - Complutense Auditory-Verbal Learning Test for Children (Test de Aprendizaje Verbal España - Complutense Infantil; TAVECI)
  - Discrimination index of word-list: False positives + omissions of recognition between 44 total words to recognize. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Verbal retention memory | 18 months
  Assessed by:
  Adults: España - Complutense Auditory-Verbal Learning Test (Test de Aprendizaje Verbal España - Complutense; TAVEC); or Infants: España - Complutense Auditory-Verbal Learning Test for Children (Test de Aprendizaje Verbal España - Complutense Infantil; TAVECI)
  - Retention index: percentatge of Long-term memory free recall between Short-term memory free recall. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Immediate visual memory | 18 months
  Assessed by: Brief Visuospatial Memory Test - Revised (BVMT-R)
  - Immediate visual memory: range: from 0 to 36. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Delayed visual memory | 18 months
  Assessed by: Brief Visuospatial Memory Test - Revised (BVMT-R)
  - Delayed visual memory: range: from 0 to 12. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Visual retention memory | 18 months
  Assessed by: Brief Visuospatial Memory Test - Revised (BVMT-R)
  - Retention index: percentatge of Long-term memory free recall between the Higher punctuation at Trial 2 or 3. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Visual recognition memory | 18 months
  Assessed by: Brief Visuospatial Memory Test - Revised (BVMT-R)
  - Figure Recognition: range: from 0 to 6. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Visual discrimination memory | 18 months
  Assessed by: Brief Visuospatial Memory Test - Revised (BVMT-R)
  - Discrimination index: figure recognized minus false positives. Range: from -6 to 6. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Processing speed | 18 months
  Processing speed Index (PSI; from Weschler Adult Intelligence Scale - IV (WAIS-IV).
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
TMT-A | 18 months
  Trail Making Test part A (TMT-A):
  - Time in seconds: from 0 to infinity.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
TMT-B | 18 months
  Trail Making Test part B (TMT-B):
  - Time in seconds: from 0 to infinity.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Naming | 18 months
  Assessed by: Boston Naming Test (BNT)
  - Total correct: from 0 to 60
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Naming with cues | 18 months
  Assessed by: Boston Naming Test (BNT)
  - Total correct with phonemic cue: from 0 to 60
Latency in naming | 18 months
  Assessed by: Boston Naming Test (BNT)
  - Time to complete test in seconds
Semantic fluency | 18 months
  Number of name of animals recalled in 1 minute: range: from 0 to infinity. (Test Barcelona - Revised) (for ADULTS) Number of name of animals recalled in 1 minute + number of name of food and drinks recalled in 1 minute: from 0 to infinity (NEPSY - II) (for CHILDREN)
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Phonemic fluency | 18 months
  Number of words started by letter "M" recalled in 1 minute: Range: from 0 to infinity. (Test Barcelona-Revised) (for ADULTS) Number of words started by letter "P" recalled in 1 minute + number of words started by letter "M" in 1 minute: range: from 0 to infinity (NEPSY-II) (for CHILDREN).
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Visuospatial skills | 18 months
  Number location subtest of the Visual-Object Spatial and Perceptual battery.
  - Range: from 0 to 10
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Visuospatial skills - children | 18 months
  Assessed by Arrows subtest of NEPSY-2 battery
  - Range: from 0 to 20
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Stroop test - word subtest | 18 months
  - Words: words read in 45 seconds
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Stroop test - color subtest | 18 months
  - Colour: colours distinguished in 45 seconds.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Stroop test - word-color subtest | 18 months
  - Word-colour: colours distinguished in 45 seconds.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Detectability - CPT3 | 18 months
  Assessed by Continuous Performance Test - 3rd Version.
  Measures the respondent's ability to differentiate non-targets (i.e. the letter X) from targets (i.e. all other letters).
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Omissions - CPT3 | 18 months
  Assessed by Continuous Performance Test - 3rd Version.
  Result from a failure to respond to targets.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Comissions - CPT3 | 18 months
  Assessed by Continuous Performance Test - 3rd Version.
  Comissions are made when responses are given to non-targets.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
HRT - CPT3 | 18 months
  Assessed by Continuous Performance Test - 3rd Version.
  Hit Reaction Time (HRT) is the mean response speed of correct responses from the whole administration.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
HRT-SD - CPT3 | 18 months
  Assessed by Continuous Performance Test - 3rd Version.
  Hit Reaction Time Standard Deviation (HRT-SD) is a measure of response speed consistency during the entire administration.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Variability- CPT3 | 18 months
  Assessed by Continuous Performance Test - 3rd Version.
  The amount of variability that the patient showed in 18 separate segments of the administration in relation to their own overall Hit Reaction Time Standard Deviation (HRT-SD).
  It is a measure of response consistency and a "within respondent" measure".
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
HRT Block Change - CPT3 | 18 months
  Assessed by Continuous Performance Test - 3rd Version.
  Hit Reaction Time Block Change indicates the change in mean response speed across blocks.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
HRT ISI Change - CPT3 | 18 months
  Assessed by Continuous Performance Test - 3rd Version.
  Hit Reaction Time Inter-Stimulus Interval Change (HRT ISI Change) indicates the change in mean response speed at various ISIs.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Prensence of psychiatric symptoms or disorders in presential assessments | 18 months
  Number of participants with psychiatric symptoms/disorders following DSM-IV-TR guidelines (psychotic symptoms, symptoms of depression, symptoms of mania, global functioning).
Sleep microstructure - Total study time | 18 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Total sleep time: minutes
Sleep microstructure - Total sleep time | 18 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Total sleep time: minutes
Sleep microstructure - Sleep efficiency | 18 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Sleep efficiency: based on total study time and total sleep time
Sleep microstructure - Time to sleep onset | 18 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Time to sleep onset: minutes
Sleep microstructure - Time in stage N1 | 18 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Time in stage N1: minutes
Sleep microstructure - Time in stage N2 | 18 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Time in stage N2: minutes
Sleep microstructure - Time in stage N3 | 18 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Time in stage N3: minutes
Sleep microstructure - Time in stage R | 18 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Time in stage R: minutes
Sleep microstructure - First epoch of N1 | 18 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - First epoch of N1: minutes
Sleep microstructure - First epoch of N2 | 18 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - First epoch of N2: minutes
Sleep microstructure - First epoch of N3 | 18 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - First epoch of N3: minutes
Sleep microstructure - First epoch of REM | 18 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - First epoch of REM: minutes
Sleep microstructure - REM/NREM time ratio | 18 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - REM/NREM time ratio
Sleep microstructure - Number of arousals | 18 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Number of arousals (total)
Sleep microstructure - Arousal Index | 18 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Arousal Index
Sleep microstructure - Confusional arousals | 18 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Confusional arousals: Yes or No
Sleep microstructure - Direct transition from N3 to W | 18 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Direct transition from N3 to W: yes or no
Sleep microstructure - Delta arousals | 18 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - "Delta arousals"?: yes, no or unknown
Sleep microstructure - Wake after sleep | 18 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Wake after sleep: hour
Adherence to cognitive treatment - 6 months | 6 months
  Number of sessions performed in 6 months
Adherence to cognitive treatment - 9 months | 9 months
  Number of sessions performed in 9 months
Adherence to cognitive treatment - 12 months | 12 months
  Number of sessions performed in 12 months

SECONDARY OUTCOMES:
Immune/inflammatory signaling-target gene expression pathways | 18 months
  Whole blood/CSF will be collected using PAXgene® Blood RNA Tubes (Qiagen) shipped to the centers. Blood from healthy subjects and CSF from patients with normal pressure hydrocephalus will serve as controls.
  Total RNA will be extracted using PAXgene® Blood RNA Kit (Qiagen). RNA samples are quantified using Qubit 2.0 Fluorometer (Life Technologies) and RNA integrity is determined with Agilent 2100 Bioanalyzer (Agilent Technologies).
  Expression levels of 44 genes related to immune/inflammatory (or cytokine) pathways will be measured with the nCounter® Digital Analyzer (NanoString).
  The raw copy number of mRNA transcripts of each gene will be standardized (stdGene) using the geometric mean of the 4 housekeeping genes for each subject.
Neurofilament light chain (NfL) levels in acute stage | 18 months
  Signature of molecular biomarkers in the acute stage
Neurofilament light chain (NfL) levels in post-acute stage | 18 months
  Signature of molecular biomarkers in the post-acute stages
Cell immunophenotyping - proportion of CD4 | 18 months
  Whole blood/CSF obtained in a EDTA tube will be analyzed in a FACS Canto II cytometer to assess the proportion of CD4.
Cell immunophenotyping - proportion of CD8 | 18 months
  Whole blood/CSF obtained in a EDTA tube will be analyzed in a FACS Canto II cytometer to assess the proportion of CD8.
Cell immunophenotyping - proportion of CD8+CD45RA+ | 18 months
  Whole blood/CSF obtained in a EDTA tube will be analyzed in a FACS Canto II cytometer to assess the proportion of CD8+CD45RA+.
Cell immunophenotyping - proportion of CD8+CD45RO+ | 18 months
  Whole blood/CSF obtained in a EDTA tube will be analyzed in a FACS Canto II cytometer to assess the proportion of CD8+CD45RO+.
Cell immunophenotyping - proportion of iNKT | 18 months
  Whole blood/CSF obtained in a EDTA tube will be analyzed in a FACS Canto II cytometer to assess the proportion of iNKT.
Cell immunophenotyping - proportion of CD19 | 18 months
  Whole blood/CSF obtained in a EDTA tube will be analyzed in a FACS Canto II cytometer to assess the proportion of CD19.
Cell immunophenotyping - proportion of B naive (IgM+IgD+CD27-) | 18 months
  Whole blood/CSF obtained in a EDTA tube will be analyzed in a FACS Canto II cytometer to assess the proportion of B naive (IgM+IgD+CD27-).
Cell immunophenotyping - proportion of B memory (IgD-) | 18 months
  Whole blood/CSF obtained in a EDTA tube will be analyzed in a FACS Canto II cytometer to assess the proportion of B memory (IgD-).
Cell immunophenotyping - proportion of regulatory B cells | 18 months
  Whole blood/CSF obtained in a EDTA tube will be analyzed in a FACS Canto II cytometer to assess the proportion of regulatory B cells.
Cell immunophenotyping - proportion of plasmablasts | 18 months
  Whole blood/CSF obtained in a EDTA tube will be analyzed in a FACS Canto II cytometer to assess the proportion of plasmablasts.
Cell immunophenotyping - proportion of NK cells | 18 months
  Whole blood/CSF obtained in a EDTA tube will be analyzed in a FACS Canto II cytometer to assess the proportion of NK cells.
MRI | 18 months
  It will be conducted on a 3 Tesla Prisma scanner using a 32-channel head coil. Scanning takes ~50 min including 3D T1-weighted in sagittal plane; T2*axial EPI; axial diffusion weighted EPI; 3D sagittal FLAIR; resting state functional MRI and glutamate and H2O univoxel spectroscopy in dorsolateral prefrontal cortex and hippocampus. There is no contrast used for the MRI scans
  Outcome for MRI is normal or abnormal. Investigators will review all MRI sequences and determine if the MRI is abnormal and then describe the abnormality or abnormalities seen.
EEG: normalcy | 18 months
  It will include standard clinical EEG protocol (43 channels, 512 Hz18) (primary variables), and EEG reactivations of memories prior to new trials (secondary variables) while participants perform WM tasks, which will be synchronized with the task software in a laptop. The memory content from alpha power across electrodes will be related to the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Performances of the subjects produces a reactivation of memory prior to new trials while participants perform working memory tasks, and relate the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  - Normalcy: yes or no.
EEG: time awake | 18 months
  It will include standard clinical EEG protocol (43 channels, 512 Hz18) (primary variables), and EEG reactivations of memories prior to new trials (secondary variables) while participants perform WM tasks, which will be synchronized with the task software in a laptop. The memory content from alpha power across electrodes will be related to the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Performances of the subjects produces a reactivation of memory prior to new trials while participants perform working memory tasks, and relate the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Parameters:
  - Time awake: percentage
EEG: time in drowsiness | 18 months
  It will include standard clinical EEG protocol (43 channels, 512 Hz18) (primary variables), and EEG reactivations of memories prior to new trials (secondary variables) while participants perform WM tasks, which will be synchronized with the task software in a laptop. The memory content from alpha power across electrodes will be related to the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Performances of the subjects produces a reactivation of memory prior to new trials while participants perform working memory tasks, and relate the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Parameters:
  - Time in drowsiness: percentage
EEG: time asleep | 18 months
  It will include standard clinical EEG protocol (43 channels, 512 Hz18) (primary variables), and EEG reactivations of memories prior to new trials (secondary variables) while participants perform WM tasks, which will be synchronized with the task software in a laptop. The memory content from alpha power across electrodes will be related to the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Performances of the subjects produces a reactivation of memory prior to new trials while participants perform working memory tasks, and relate the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Parameters:
  - Time asleep: percentage
EEG: epileptiform activity | 18 months
  It will include standard clinical EEG protocol (43 channels, 512 Hz18) (primary variables), and EEG reactivations of memories prior to new trials (secondary variables) while participants perform WM tasks, which will be synchronized with the task software in a laptop. The memory content from alpha power across electrodes will be related to the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Performances of the subjects produces a reactivation of memory prior to new trials while participants perform working memory tasks, and relate the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Parameters:
  - Epileptiform activity: yes or no
EEG: seizures | 18 months
  It will include standard clinical EEG protocol (43 channels, 512 Hz18) (primary variables), and EEG reactivations of memories prior to new trials (secondary variables) while participants perform WM tasks, which will be synchronized with the task software in a laptop. The memory content from alpha power across electrodes will be related to the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Performances of the subjects produces a reactivation of memory prior to new trials while participants perform working memory tasks, and relate the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Parameters:
  - Seizures: yes or no
EEG: slowing | 18 months
  It will include standard clinical EEG protocol (43 channels, 512 Hz18) (primary variables), and EEG reactivations of memories prior to new trials (secondary variables) while participants perform WM tasks, which will be synchronized with the task software in a laptop. The memory content from alpha power across electrodes will be related to the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Performances of the subjects produces a reactivation of memory prior to new trials while participants perform working memory tasks, and relate the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Parameters:
  - EEG slowing: yes or no
EEG: Changes with Intermittent Light Stimulation | 18 months
  It will include standard clinical EEG protocol (43 channels, 512 Hz18) (primary variables), and EEG reactivations of memories prior to new trials (secondary variables) while participants perform WM tasks, which will be synchronized with the task software in a laptop. The memory content from alpha power across electrodes will be related to the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Performances of the subjects produces a reactivation of memory prior to new trials while participants perform working memory tasks, and relate the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Parameters:
  - Changes with Intermittent Light Stimulation: yes or no
EEG: Changes with hyperventilation | 18 months
  It will include standard clinical EEG protocol (43 channels, 512 Hz18) (primary variables), and EEG reactivations of memories prior to new trials (secondary variables) while participants perform WM tasks, which will be synchronized with the task software in a laptop. The memory content from alpha power across electrodes will be related to the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Performances of the subjects produces a reactivation of memory prior to new trials while participants perform working memory tasks, and relate the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Parameters:
  - Changes with hyperventilation: yes or no
Verbal working memory - remote assessment | 18 months
  Assessed by:
  Digit subtest from WAIS-IV: obtained by Forward order, indirect order, increasing order subtests.
  - Range: 0 - 48
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Verbal learning - remote assessment | 18 months
  Assessed by:
  Total learning List A subtest from Rey Auditory Verbal Learning Test (RAVLT)
  - Range: 0 - 75
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Proactive interference verbal memory - remote assessment | 18 months
  Assessed by:
  List B subtest from Rey Auditory Verbal Learning Test (RAVLT)
  - Range: 0 - 15
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Short-term verbal memory - remote assessment | 18 months
  Assessed by:
  Short-term verbal memory subtest from Rey Auditory Verbal Learning Test (RAVLT)
  - Range: 0 - 15
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Long-term verbal memory - remote assessment | 18 months
  Assessed by:
  Long-term verbal memory subtest from Rey Auditory Verbal Learning Test (RAVLT)
  - Range: 0 - 15
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Verbal recognition memory - remote assessment | 18 months
  Assessed by:
  Verbal recognition memory list subtest from Rey Auditory Verbal Learning Test (RAVLT)
  - Range: 0 - 15
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Verbal discrimination memory - remote assessment | 18 months
  Assessed by:
  Verbal discrimination memory subtest from Rey Auditory Verbal Learning Test (RAVLT)
  - Range: 0 - 1
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Complex figure copy - remote assessment | 18 months
  Assessed by:
  Precision in the copy of the Rey-Osterrieth Complex Figure:
  - Range: 0-36
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Time - Complex figure copy - remote assessment | 18 months
  Assessed by:
  Time to perform the copy of the Rey-Osterrieth Complex Figure: seconds
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Type - Complex figure copy - remote assessment | 18 months
  Assessed by:
  Type of copy of the Rey-Osterrieth Complex Figure:
  - Range: 1 to 4
Short-term visual memory - remote assessment | 18 months
  Assessed by:
  Short term memory subtest of the Rey-Osterrieth Complex Figure:
  - Range: 0 - 36
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Long-term visual memory - remote assessment | 18 months
  Assessed by:
  Long-term memory subtest of the Rey-Osterrieth Complex Figure:
  - Range: 0 - 36
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Orientation in time - remote assessment | 18 months
  Assessed by:
  Orientation in time subtest from Test Barcelona - Revised.
  - Range: 0 - 5
  Higher is better.
Orientation in space - remote assessment | 18 months
  Assessed by:
  Orientation in space subtest from Test Barcelona - Revised.
  - Range: 0 -5
5DT Lecture - remote assessment | 18 months
  Assessed by:
  Lecture subtest from 5 digit test: time
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
5DT counting - remote assessment | 18 months
  Assessed by:
  Counting subtest from 5 digit test: time
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
5DT Choosing - remote assessment | 18 months
  Assessed by:
  Choosing subtest from 5 digit test: time
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
5DT Switching - remote assessment | 18 months
  Assessed by:
  Switching subtest from 5 digit test: time
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
5DT Inhibition - remote assessment | 18 months
  Assessed by:
  Inhibition subtest from 5 digit test: time
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
5DT Flexibility - remote assessment | 18 months
  Assessed by:
  Flexibility subtest from 5 digit test: time
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
IEDEEDS - remote assessment | 18 months
  IED EDS Errors: The number of times that the subject failed to select the stimulus compatible with the current rule on the stage where the extra-dimensional shift occurs. This is a measure of the subject's ability to shift attentional set.
  Assessed by:
  Intra-Extra Dimensional test from CANTAB battery.
  - Raw score range: 0 - 50. Lower is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
IEDYERTA - remote assessment | 18 months
  IED Total Errors (Adjusted): The total number of times that the subject chose a wrong stimulus - i.e. one incompatible with the current rule, adjustment for every stage that was not reached. Lower is better. Total Errors Adjusted = Total Errors (problems reached) + [(number of unreached problems) * (25)] This is a measure of the subject's efficiency in attempting the test. Subjects failing at any stage of the test will have had less opportunity to make errors. The adjustment is carried out to compensate for this missing data, and provide a more comparable error score to subjects completing all stages of the test..
  Assessed by:
  Intra-Extra Dimensional test from CANTAB battery.
  - Raw score range: 0 - 402. Lower is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
IEDYCOST - remote assessment | 18 months
  IED Stages Completed: This is the total number of stages the subject completed successfully. There are nine stages to be completed. Higher is better.
  Assessed by:
  Intra-Extra Dimensional test from CANTAB battery.
  - Range: 0 - 9. Higher is better.
SWM Total Errors - remote assessment | 18 months
  SWM Total Errors: The total number of times a box is selected that is certain not to contain a token and therefore should not have been visited by the subject, i.e. between errors + within errors - double errors. Calculated across all assessed four, six and eight token trials.
  Assessed by:
  Spatial Working Memory test from CANTAB battery.
  - Range: 0 - 157. Lower is better
SWM Between Errors - remote assessment | 18 months
  SWM Between Errors: The number of times the subject incorrectly revisits a box in which a token has previously been found. Calculated across all assessed four, six and eight token trials.
  Assessed by:
  Spatial Working Memory test from CANTAB battery:
  - Raw score range: 0 - 153. Lower is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
SWM Within Errors - remote assessment | 18 months
  SWM Within Errors: The number of times a subject revisits a box already shown to be empty during the same search. Calculated across all assessed four, six and eight token trials.
  Assessed by:
  Spatial Working Memory test from CANTAB battery:
  - Range: 0 - 153. Lower is better.
SWM Double Errors - remote assessment | 18 months
  SWM Double Errors: The number of times a subject commits an error that is both a within error and a between error. Calculated across all assessed four, six and eight token trials.
  Assessed by:
  Spatial Working Memory test from CANTAB battery:
  - Range: 0 - 147. Lower is better.
SWMS - remote assessment | 18 months
  SWM Strategy (6-8 boxes): The number of times a subject begins a new search pattern from the same box they started with previously. If they always begin a search from the same starting point we infer that the subject is employing a planned strategy for finding the tokens. Therefore a low score indicates high strategy use (1 = they always begin the search from the same box), a high score indicates that they are beginning their searches from many different boxes. Calculated across assessed trials with 6 tokens or 8 tokens.
  Assessed by:
  Spatial Working Memory test from CANTAB battery:
  - Range: 2 - 14. Lower is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased
SWMSX - remote assessment | 18 months
  SWM Strategy (6-12 boxes): The number of times a subject begins a new search pattern from the same box they started with previously. If they always begin a search from the same starting point we infer that the subject is employing a planned strategy for finding the tokens. Therefore a low score indicates high strategy use (1 = they always begin the search from the same box), a high score indicates that they are beginning their searches from many different boxes. Calculated across assessed trials with 6 tokens or more.
  Assessed by:
  Spatial Working Memory test from CANTAB battery:
  - Range: 3 - 26. Lower is better.
SWMPR - remote assessment | 18 months
  SWM Problem Reached: This measure reports the problem number that the subject reached, but did not necessarily complete.
  Assessed by:
  Spatial Working Memory test from CANTAB battery:
  - Range: 2 - 6. Higher is better.
ERTTH - remote assessment | 18 months
  Assessed by:
  Emotion Recognition Task from CANTAB battery.
  ERT Total Hits: The total number of times the subject selected the correct emotion. Calculated across all assessed trials.
  - Range: 0 - 90. Higher is Better
ERTTHH - remote assessment | 18 months
  Assessed by:
  Emotion Recognition Task from CANTAB battery.
  ERT Total Hits Happiness: The total number of times the subject correctly selected the emotion 'Happiness'. Calculated across all assessed trials.
  - Range: 0 - 15 . Higher is Better
ERTTHS - remote assessment | 18 months
  Assessed by:
  Emotion Recognition Task from CANTAB battery.
  ERT Total Hits Sadness: The total number of times the subject correctly selected the emotion 'Sadness'. Calculated across all assessed trials.
  - Range: 0 - 15 . Higher is Better
ERTTHF - remote assessment | 18 months
  Assessed by:
  Emotion Recognition Task from CANTAB battery.
  ERT Total Hits Fear: The total number of times the subject correctly selected the emotion 'Fear'. Calculated across all assessed trials.
  - Range: 0 - 15 . Higher is Better
ERTTHA - remote assessment | 18 months
  Assessed by:
  Emotion Recognition Task from CANTAB battery.
  ERT Total Hits Anger: The total number of times the subject correctly selected the emotion 'Anger'. Calculated across all assessed trials.
  - Range: 0 - 15 . Higher is Better
ERTTHSU - remote assessment | 18 months
  Assessed by:
  Emotion Recognition Task from CANTAB battery
  ERT Total Hits Surprise: The total number of times the subject correctly selected the emotion 'Surprise'. Calculated across all assessed trials.
  - Range: 0 - 15 . Higher is Better.
ERTTHD - remote assessment | 18 months
  Assessed by:
  Emotion Recognition Task from CANTAB battery.
  ERT Total Hits Disgust: The total number of times the subject correctly selected the emotion 'Disgust'. Calculated across all assessed trials.
  - Range: 0 - 15 . Higher is Better.
ERTTFAH - remote assessment | 18 months
  Assessed by:
  Emotion Recognition Task from CANTAB battery.
  ERT Total False Alarms Happiness: The total number of times the subject incorrectly selected the emotion 'Happiness'. Calculated across all assessed trials.
  - Range: 0 - 75 . Lower is Better.
ERTTFAS - remote assessment | 18 months
  Assessed by:
  Emotion Recognition Task from CANTAB battery.
  ERT Total False Alarms Sadness: The total number of times the subject incorrectly selected the emotion 'Sadness'. Calculated across all assessed trials.
  - Range: 0 - 75 . Lower is Better.
ERTTFAF - remote assessment | 18 months
  Assessed by:
  Emotion Recognition Task from CANTAB battery.
  ERT Total False Alarms Fear: The total number of times the subject incorrectly selected the emotion 'Fear'. Calculated across all assessed trials.
  - Range: 0 - 75 . Lower is Better.
ERTTFAA - remote assessment | 18 months
  Assessed by:
  Emotion Recognition Task from CANTAB battery.
  ERT Total False Alarms Anger: The total number of times the subject incorrectly selected the emotion 'Anger'. Calculated across all assessed trials.
  - Range: 0 - 75 . Lower is Better.
ERTTFASU - remote assessment | 18 months
  Assessed by:
  Emotion Recognition Task from CANTAB battery.
  ERT Total False Alarms Surprise: The total number of times the subject incorrectly selected the emotion 'Surprise'. Calculated across all assessed trials.
  - Range: 0 - 75 . Lower is Better.
ERTTFAD - remote assessment | 18 months
  Assessed by:
  Emotion Recognition Task from CANTAB battery.
  ERT Total False Alarms Disgust: The total number of times the subject incorrectly selected the emotion 'Disgust'. Calculated across all assessed trials.
  - Range: 0 - 75 . Lower is Better.
ERTUHRH - remote assessment | 18 months
  Assessed by:
  Emotion Recognition Task from CANTAB battery.
  ERT Unbiased Hit Rate Happiness: The unbiased hit rate ensures that recognition accuracy of the Happiness emotion is not influenced by response guessing or response bias effects. It takes into consideration the joint probability of an individual making a correct response, based on the presentation of the correct stimulus out of the available possibilities. Calculated for assessed Happiness trials only.
  - Range: 0 to 1. Higher is better.
ERTUHRS - remote assessment | 18 months
  Assessed by:
  Emotion Recognition Task from CANTAB battery.
  ERT Unbiased Hit Rate Sadness: The unbiased hit rate ensures that recognition accuracy of the Sadness emotion is not influenced by response guessing or response bias effects. It takes into consideration the joint probability of an individual making a correct response, based on the presentation of the correct stimulus out of the available possibilities. Calculated for assessed Sadness trials only
  - Range: 0 to 1. Higher is better.
ERTUHRF - remote assessment | 18 months
  Assessed by:
  Emotion Recognition Task from CANTAB battery.
  ERT Unbiased Hit Rate Fear: The unbiased hit rate ensures that recognition accuracy of the Fear emotion is not influenced by response guessing or response bias effects. It takes into consideration the joint probability of an individual making a correct response, based on the presentation of the correct stimulus out of the available possibilities. Calculated for assessed Fear trials only.
  - Range: 0 to 1. Higher is better.
ERTUHRA - remote assessment | 18 months
  Assessed by:
  Emotion Recognition Task from CANTAB battery.
  ERT Unbiased Hit Rate Anger: The unbiased hit rate ensures that recognition accuracy of the Anger emotion is not influenced by response guessing or response bias effects. It takes into consideration the joint probability of an individual making a correct response, based on the presentation of the correct stimulus out of the available possibilities. Calculated for assessed Anger trials only.
  - Range: 0 to 1. Higher is better.
ERTUHRSU - remote assessment | 18 months
  Assessed by:
  Emotion Recognition Task from CANTAB battery.
  ERT Unbiased Hit Rate Surprise: The unbiased hit rate ensures that recognition accuracy of the Surprise emotion is not influenced by response guessing or response bias effects. It takes into consideration the joint probability of an individual making a correct response, based on the presentation of the correct stimulus out of the available possibilities. Calculated for assessed Anger trials only.
  - Range: 0 to 1. Higher is better.
ERTUHRSD - remote assessment | 18 months
  Assessed by:
  Emotion Recognition Task from CANTAB battery.
  ERT Unbiased Hit Rate Disgust: The unbiased hit rate ensures that recognition accuracy of the Disgust emotion is not influenced by response guessing or response bias effects. It takes into consideration the joint probability of an individual making a correct response, based on the presentation of the correct stimulus out of the available possibilities. Calculated for assessed Disgust trials only.
  - Range: 0 to 1. Higher is better.
Semantic fluency - remote assessment | 18 months
  Assessed by:
  Semantic fluency test:
  * Produce names of fruits and vegetables in 1 minute (Test Barcelona - Revised) (for ADULTS)
  * Number of name of animals recalled in 1 minute + number of name of food and drinks recalled in 1 minute: from 0 to infinity (NEPSY - II) (for CHILDREN)
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Phonemic fluency - remote assessment | 18 months
  Assessed by:
  Phonemic fluenct test:
  * Produce words that start with letter M in 1 minute: range from 0 to infinity (Test Barcelona - Revised) (for ADULTS)
  * Number of words started by letter "P" recalled in 1 minute + number of words started by letter "M" in 1 minute: range: from 0 to infinity (NEPSY-II) (for CHILDREN).
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Naming - remote assessment | 18 months
  Assessed by:
  Boston Naming Test (BNT):
  - Range: from 0 to 60
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Naming with cues - remote assessment | 18 months
  Assessed by: Boston Naming Test (BNT)
  - Total correct with phonemic cue: from 0 to 60
Time in Naming - remote assessment | 18 months
  Assessed by: Boston Naming Test (BNT): time to complete
Visuospatial skills - remote assessment | 18 months
  Assessed by:
  Benton Judgment of Line Orientation Test (JLO):
  - Range: 0 to 30
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Psychiatric symptoms/disorders in remote assessments | 18 months
  Number of participants with psychiatric symptoms/disorders following DSM-IV-TR guidelines (psychotic symptoms, symptoms of depression, symptoms of mania, global functioning).
Serial bias in working memory | 18 months
  This is quantified from the participant responses in the working memory task. Errors in the report of memorized locations are multiplied by the sign of the difference in locations in the previous and current trials and then averaged over the whole session to obtain the index of serial bias. We expect increases in this index as patients improve clinically.
EEG reactivations in working memory | 18 months
  This is quantified by training decoders of memorized locations on EEG signals acquired over several electrodes during the working memory task. Reactivations are the average strength of the decoders during the fixation period of the next trial. We expect that EEG reactivations increase as patients improve clinically and correlate with the serial bias index.
Slow-wave rate of growth during slow-wave sleep period | 18 months
  This is quantified from EEG recorded during sleep, by detecting individual slow-waves and estimating their strength, and then computing the rate of growth of this strength in the first slow-wave periods in the night. We expect the rate of growth of slow waves to increase as patients improve.

CONTACTS AND LOCATIONS:
Overall Officials: Josep Dalmau, MD, PhD, Principal Investigator — Hospital Clínic
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Catalonia, Spain

REFERENCES:
- [Background] Guasp M, Rosa-Justicia M, Munoz-Lopetegi A, Martinez-Hernandez E, Armangue T, Sugranyes G, Stein H, Borras R, Prades L, Arino H, Planaguma J, De-La-Serna E, Escudero D, Llufriu S, Sanchez-Valle R, Santamaria J, Compte A, Castro-Fornieles J, Dalmau J; Spanish anti-NMDAR Encephalitis Study Group. Clinical characterisation of patients in the post-acute stage of anti-NMDA receptor encephalitis: a prospective cohort study and comparison with patients with schizophrenia spectrum disorders. Lancet Neurol. 2022 Oct;21(10):899-910. doi: 10.1016/S1474-4422(22)00299-X. PMID 36115362
- [Background] Titulaer MJ, McCracken L, Gabilondo I, Armangue T, Glaser C, Iizuka T, Honig LS, Benseler SM, Kawachi I, Martinez-Hernandez E, Aguilar E, Gresa-Arribas N, Ryan-Florance N, Torrents A, Saiz A, Rosenfeld MR, Balice-Gordon R, Graus F, Dalmau J. Treatment and prognostic factors for long-term outcome in patients with anti-NMDA receptor encephalitis: an observational cohort study. Lancet Neurol. 2013 Feb;12(2):157-65. doi: 10.1016/S1474-4422(12)70310-1. Epub 2013 Jan 3. PMID 23290630
- [Background] Arino H, Munoz-Lopetegi A, Martinez-Hernandez E, Armangue T, Rosa-Justicia M, Escudero D, Matos N, Graus F, Sugranyes G, Castro-Fornieles J, Compte A, Dalmau J, Santamaria J. Sleep disorders in anti-NMDAR encephalitis. Neurology. 2020 Aug 11;95(6):e671-e684. doi: 10.1212/WNL.0000000000009987. Epub 2020 Jun 23. PMID 32576635
- [Background] Finke C, Kopp UA, Scheel M, Pech LM, Soemmer C, Schlichting J, Leypoldt F, Brandt AU, Wuerfel J, Probst C, Ploner CJ, Pruss H, Paul F. Functional and structural brain changes in anti-N-methyl-D-aspartate receptor encephalitis. Ann Neurol. 2013 Aug;74(2):284-96. doi: 10.1002/ana.23932. Epub 2013 Jul 8. PMID 23686722
- [Background] Heine J, Kopp UA, Klag J, Ploner CJ, Pruss H, Finke C. Long-Term Cognitive Outcome in Anti-N-Methyl-D-Aspartate Receptor Encephalitis. Ann Neurol. 2021 Dec;90(6):949-961. doi: 10.1002/ana.26241. Epub 2021 Oct 21. PMID 34595771
- [Background] Armangue T, Titulaer MJ, Malaga I, Bataller L, Gabilondo I, Graus F, Dalmau J; Spanish Anti-N-methyl-D-Aspartate Receptor (NMDAR) Encephalitis Work Group. Pediatric anti-N-methyl-D-aspartate receptor encephalitis-clinical analysis and novel findings in a series of 20 patients. J Pediatr. 2013 Apr;162(4):850-856.e2. doi: 10.1016/j.jpeds.2012.10.011. Epub 2012 Nov 16. PMID 23164315

DOCUMENTS (5):
  • Study Protocol (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/88/NCT06183788/Prot_000.pdf
  • Informed Consent Form: IC for adult patients (2022-12-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT06183788/ICF_001.pdf
  • Informed Consent Form: IC for adult familiar (2022-12-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT06183788/ICF_002.pdf
  • Informed Consent Form: IC for minors/patients under the age of 18 (2022-12-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT06183788/ICF_003.pdf
  • Informed Consent Form: IC for familiar of minors/patients under the age of 18 (2022-12-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT06183788/ICF_004.pdf